CLINICAL TRIAL: NCT05731570
Title: Cognitive Impairment in Long Covid: PhEnotyping and RehabilitatiOn (CICERO)
Brief Title: Cognitive Rehabilitation for People With Cognitive Covid19
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Bangor University (Other); St George's University Hospitals NHS Foundation Trust (Other); University of Brighton (Other); University Hospital Southampton NHS Foundation Trust (Other); Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICERO clinical trial
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Long Covid19
Keywords: cognitive rehabilitation; brain fog; Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; COVID-19 | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): cognitive rehabilitation programme. 1h session per week x 10 weeks
  Interventions: Behavioral: Cognitive rehabilitation
- Control (No Intervention): The control group receives treatment as usual, this is, participants will carry on with the care they were receiving prior to entry in the study.

INTERVENTIONS:
Behavioral: Cognitive rehabilitation — Set of restorative and compensatory strategies to rehabilitate cognitive function combined with emotional regulation techniques.
  Arms: Intervention

SUMMARY:
Cognitive impairment is increasingly recognised as a major component of long Covid, and is estimated to be present in 25-75% of affected individuals. This impairment impacts quality of life and the loss of functional ability has major consequences for affected people, their families and the wider economy given people's difficulty in returning to work.

This study will focus on helping people recover from cognitive Covid. This will involve use of rehabilitation strategies aimed at improving function in those cognitive functions identified in Stage 1 as being most affected, and assessing the benefit of rehabilitation on quality of life and people's ability to return to everyday function. These strategies will be co-produced in collaboration with a group of people living with cognitive Covid. At the end of Stage 2 we will produce a freely available "Covid-19 Cognitive Recovery Guide" for affected people, their close contacts and clinicians.

In conclusion, cognitive impairment is frequently observed in long Covid but at present little is understood about its nature, or how it can be treated. The sheer scale of the CV19 pandemic makes this a top priority unmet need for healthcare worldwide. The aim of this study is to meet this need and to deliver a treatment plan for affected people which will help them return to normal life and working ability.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 30 and 60 years
2. Evidence of prior CV19 infection:

   * either positive CV19 PCR
   * or positive CV19 antibody test
   * or acute symptoms consistent with the recognised core features of acute CV19 infection and post-acute symptoms consistent with the recognised core features of long Covid
3. Cognitive impairment persisting more than three months after the acute CV19 infection, defined in terms of subjective reports of cognitive decline post-infection

Exclusion Criteria:

1. Cognitive impairment prior to CV19 infection
2. Occurrence of acute neurological disorder, such as stroke or encephalitis, that could give rise to cognitive sequelae
3. People who are on any medications that are considered by the study investigators to have significant adverse effects on cognition
4. A pre-existing major psychiatric or medical disorder that is considered by the study investigators to have potential to affect cognition
5. High alcohol intake
6. Recreational drug use
7. Loss of mental capacity such that the affected individual is unable to give informed consent
8. Participants will not be eligible for Workstream 2 if they do not exhibit significant impairment on baseline cognitive assessments, as they will not gain from cognitive rehabilitation.
9. Participants with pacemakers or other implanted devices, those with metal foreign bodies (e.g. shrapnel from war injuries) and those who have had certain types of surgery will be excluded from the MRI substudy. Although MRI is not known to affect the unborn child, we will also exclude subjects who may be pregnant just to be on the safe side.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Goal-attainment | measured at baseline, 3 and 6 months post-randomisation
  performance on goals selected by participants

SECONDARY OUTCOMES:
Change in cognitive function | measured at baseline, 3 and 6 months post-randomisation
  set of tests to measure objective improvements in cognitive function
Change in quality of life (EQ-5D-5L) | measured at baseline, 3 and 6 months post-randomisation
  Measure of quality of life
Change in Life Space Questionnaire | measured at baseline, 3 and 6 months post-randomisation
  Measures the extent of mobility
Social Functioning (SF-DEM) | measured at baseline, 3 and 6 months post-randomisation
  patient reported outcome measure to assess social functioning
Change in Instrumental Activities of Daily Living (IADL) Scale | measured at baseline, 3 and 6 months post-randomisation
  assessment of independent living skills
Generalised Anxiety Disorder Assessment (GAD-7) | measured at baseline, 3 and 6 months post-randomisation
  measures levels of anxiety
Change in Patient Health Questionnaire (PHQ-8) | measured at baseline, 3 and 6 months post-randomisation
  measures depressive disorders
Change in Chalder Fatigue Scale | measured at baseline, 3 and 6 months post-randomisation
  measures the severity of tiredness in fatiguing illnesses
Change in Pittsburgh Sleep Quality (PSQI) | measured at baseline, 3 and 6 months post-randomisation
  slef reported questionnaire that assesses sleep quality
Change in DePaul Symptom Questionnaire - Post-Exertional Malaise (DSQ-PEM). | measured at baseline, 3 and 6 months post-randomisation
  measures presence and severity of post-exertional malaise
Change in Client Service Receipt Inventory (CSRI) | measured at baseline, 3 and 6 months post-randomisation
  tool used to collect information on the whole range of services and supports study participants may use

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chan, Dr, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanova M, Patel AMR, Scott I, Gilpin G, Manning EN, Ash C, Wittenberg P, Lim J, Hoare Z, Evans R, Bray N, Kipps CM, Devine C, Ahmed S, Dunne R, Koniotes A, Warren C, Chan D, Suarez-Gonzalez A. Telehealth-delivered cognitive rehabilitation for people with cognitive impairment as part of the post-COVID syndrome: protocol for a randomised controlled trial as part of the CICERO (Cognitive Impairment in Long COVID: Phenotyping and Rehabilitation) study. Trials. 2024 Oct 22;25(1):704. doi: 10.1186/s13063-024-08554-3. PMID 39434179